CLINICAL TRIAL: NCT05021848
Title: Effects of a Partnered Multicomponent Exercise Program on Improving the Physical Function and Well-being of Elderly People in Long-term Care Facilities
Brief Title: Partnered Multicomponent Exercise for Elderly in Long-term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, CY Song, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-046-B
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Exercise; Long Term Care Facilities; Physical Function; Happiness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group (N=14) received a 90-minute partnered multicomponent exercises intervention once weekly for 12 weeks
  Interventions: Other: partnered multicomponent exercises program
- control group (No Intervention): The control group (N=14) carried out the usual activities without intervention. (After 12-wk, multicomponent exercises intervention will be given)

INTERVENTIONS:
Other: partnered multicomponent exercises program — aerobic,strength, flexibility and balance exercises and game
  Arms: Experimental group

SUMMARY:
This study aimed to explore the effects of a partnered multicomponent exercise program on improving the physical function and sense of well-being of elderly people in Long-term Care Facilities (LTCFs).

DETAILED DESCRIPTION:
This study is a single-blinded randomized controlled trial. Elderly residents were recruited from two LTCFs in Yilan county. The experimental group (N=14) received a 90-minute partnered multicomponent exercises intervention once weekly for 12 weeks. The control group (N=14) carried out the usual activities without intervention. The Barthel Index (BI), Short Physical Performance Battery (SPPB), De Morton Mobility Index(DEMMI), handgrip strength, and Chinese Happiness Inventory (CHI) were measured before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Over 60years old,living in the long term care facilities,after Physician agrees.No infectious diseases.

Exclusion Criteria:

1. Acute disease or unstable state (such as heart failure).
2. Severe musculoskeletal diseases (such as fractures, lower limb joint pain and deformation).
3. Cognitive impairment (MMSE<20) .
4. At the end of life.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change of activities of daily living function | before , after 12-weeks interventions
  Barthel Index (BI)
Change of physical function | before , after 12-weeks interventions
  Short Physical Performance Battery (SPPB)
Change of mobility | before , after 12-weeks interventions
  de Morton Mobility Index(DEMMI)
Change of grip strength | before , after 12-weeks interventions
  Handgrip strength
Change of sense of well-being | before , after 12-weeks interventions
  Chinese Happiness Inventory (CHI)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Yi Song, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided